CLINICAL TRIAL: NCT01259388
Title: A Pilot Trial of Lithium in Progressive Multiple Sclerosis
Brief Title: A Pilot Study of Lithium in Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CDA2-003-10S
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Lithium
MeSH Terms: conditions — Multiple Sclerosis | interventions — Lithium Carbonate; Standard of Care; Observation

STUDY DESIGN:
Intervention Model Description: Each study participant agreed to a two-year enrollment commitment. Each subject was asked to take lithium for one year and to be observed for one year. Randomization was used to determine the sequence of lithium vs. observation (year 1 or year 2).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium (Experimental): Lithium-treatment phase
  Lithium Carbonate: Lithium carbonate is dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time.
  Interventions: Drug: Lithium Carbonate
- Observation (No Intervention): During observation subjects continue on their standard of care disease modifying agent (or no agent at all if judged not appropriate by the treating physician).

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium carbonate is dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time.
  Other Names: Standard care (observation)
  Arms: Lithium

SUMMARY:
The purpose of this study is to determine whether lithium carbonate is safe, well-tolerated, and effective at treating progressive forms of multiple sclerosis.

DETAILED DESCRIPTION:
In progressive multiple sclerosis (MS), patients experience worsening disability through a combination of inflammatory and neuro-degenerative processes. To test whether low-dose lithium carbonate ameliorates disability accumulation in progressive MS, patients with progressive MS were randomly assigned to take lithium in either the first or second year of a two-year trial. The trial was designed as a cross-over study to maximize exposure to lithium to for two reasons: 1) To increase the number of persons with MS exposed to lithium for purposes of assessing safety and tolerance; and 2) To increase the power to detect changes in the primary radiological outcome (change in brain volume) and also in secondary clinical outcomes (disability, mood, fatigue, cognition).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a progressive subtype of multiple sclerosis by revised 2005 McDonald Criteria.
* EDSS of 3.0-6.5
* Ages 30-65
* Must be mentally capable of providing informed consent and following study guidelines.

Exclusion Criteria:

* Relapse or steroid treatment within 1 month of trial entry.
* Any current or previous treatment with mitoxantrone, azathioprine, methotrexate, mycophenolate, cyclophosphamide, or any experimental therapy.
* Women who are pregnant, wishing to become pregnant in the coming 30 months, or are breastfeeding.
* Sexually active women unwilling to use reliable contraception (oral contraceptives, condom, IUD).
* Patients with known kidney dysfunction or creatinine >1.4; known cardiac arrhythmia or significant conduction abnormality on EKG; uncontrolled thyroid disease or TSH >20% above the upper limit of normal; uncontrolled psoriasis, HIV, or any other severe medical condition.
* Patients with a history of unstable psychiatric illness or active severe depression.
* Patients with a history of seizure.
* Concurrent use of any of the following medications: Antipsychotics, diuretics, digoxin, or iodide salts.
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) 5 or more days a week.
* Patients with a history of substance abuse in the past year.
* Patients sensitive to gadolinium, or who are unable to undergo the required number of MRI scans.
* Unable to speak or understand sufficient English to consent or complete study procedures.
* Patients unable or unwilling to provide informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Rinker, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Kirklin Clinic, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinker JR 2nd, Meador WR, King P. Randomized feasibility trial to assess tolerance and clinical effects of lithium in progressive multiple sclerosis. Heliyon. 2020 Jul 28;6(7):e04528. doi: 10.1016/j.heliyon.2020.e04528. eCollection 2020 Jul. PMID 32760832

RESULTS

PARTICIPANT FLOW:
Groups:
- Lithium First (One Year), Then Observation (One Year): Subjects randomized to this group took lithium carbonate dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time, followed by a year of observation (standard care). No washout period occurred between the treatment periods.
- Observation First (One Year), Then Lithium (One Year): Subjects randomized to this group were observed for a year of observation (standard care), followed by a year of lithium carbonate dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time. No washout period occurred between the treatment periods.
Period: Overall Study
Arm/Group | Lithium First (One Year), Then Observation (One Year) | Observation First (One Year), Then Lithium (One Year)
Started | 11 | 12
Completed | 6 | 11
Not Completed | 5 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lithium Then Observation: Lithium carbonate was dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time.
  During observation subjects continued on their standard of care disease modifying agent (or no agent at all if judged not appropriate by the treating physician).
- Observation Then Lithium: During observation subjects continued on their standard of care disease modifying agent (or no agent at all if judged not appropriate by the treating physician).
  Lithium carbonate was dosed at 150 or 300 mg daily, as tolerated by study subjects, for one year's time.
- Total: Total of all reporting groups
Arm/Group | Lithium Then Observation | Observation Then Lithium | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (4.6) | 47.1 (8.1) | 51.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Brain Parenchymal Fraction
Description: Paired comparison of change in brain parenchymal fraction during Lithium treatment and during observation period
Time Frame: 2 years
Population: Due to this being a crossover study design, each participant's data was evaluated for each phase of the trial (Li treatment and observation). Only subjects who completed both years (and thus both phases) of the study were included.
Measure: Mean (Standard Error); unit: percentage of change in brain volume
Groups:
- Observation: During observation subjects continued on their standard of care disease modifying agent (or no agent at all if judged not appropriate by the treating physician).
Arm/Group | Lithium | Observation
Number analyzed (Participants) | 17 | 17
percentage of change in brain volume | 0.107 (0.38) | -0.355 (0.22)
Statistical Analysis 1: Comparison: Lithium vs Observation; Test type: Superiority or Other; p = 0.346, t-test, 2 sided

2. Secondary Outcome: Total Relapses
Description: Total number of relapses which occurred during the Li-treatment and observation study phases.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: relapses
Arm/Group | Lithium | Observation
Number analyzed (Participants) | 17 | 17
relapses | 2 | 5

3. Secondary Outcome: Change in Expanded Disability Status Scale Score
Description: The Expanded Disability Status Scale (EDSS) is an ordinal scale ranging from 0 to 10 used to assess disability in multiple sclerosis (MS). A score of 0 denotes no neurological impairments and no neurological exam abnormalities, while a score of 10 denotes death due to MS. The EDSS is derived from subscales called Functional System Scales at the lower range of the EDSS, and from ambulatory impairments and overall functional impairment at higher ranges of the scale. The Functional System scores (Vision, Brainstem, Pyramidal, Sensory, Cerebellar, Cognitive, Bladder and Bowel) are used to generate the EDSS based on pre-specified rules that determine the overall EDSS score.
Time Frame: 2 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Lithium | Observation
Number analyzed (Participants) | 17 | 17
Units on a scale | 0 [0 to 0] | 0.5 [0 to 1]
Statistical Analysis 1: Comparison: Lithium vs Observation; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire period of study involvement (2 years). For each subject, 1 year was observation and the other year subjects were taking the study medication, lithium carbonate.
Description: Serious and unexpected adverse events were collected for both lithium and observation years. However, since this was an open-label study, subjects were only asked about medication side effects during the lithium-treatment portion of the study. For this reason the Observation period does not list non-serious adverse events.
Arm/Group | Lithium | Observation
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/18
Other Adverse Events (participants affected / at risk) | 22/23 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lithium (N=23) | Observation (N=18)
Hospitalization to place suprapubic catheter (Renal and urinary disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=23) | Observation (N=18)
Excess thirst (General disorders) | 18 (112) | 0
Fatigue (General disorders) | 15 | 0
Polyuria (Renal and urinary disorders) | 15 | 0
Weight gain (General disorders) | 13 | 0
Weight loss (General disorders) | 10 | 0
Tremor (Nervous system disorders) | 10 | 0
Cognitive change (Nervous system disorders) | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 0
Gait impairment (Nervous system disorders) | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 0
Increased TSH (Endocrine disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Unusual dreams (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This was a pilot study and thus by design was not powered to detect therapeutic differences. The primary purpose of the study was feasibility with the specified outcomes intended to generate preliminary data for subsequent research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes